CLINICAL TRIAL: NCT00991822
Title: A Double-masked Comparison of the Effect of Dorzolamide and Timolol on Optic Disk Blood Flow in Patients With Open Angle Glaucoma
Brief Title: A Comparison of the Effect of Dorzolamide and Timolol on Optic Disk Blood Flow in Patients With Open Angle Glaucoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: HG Eichler, MD, Prof, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OPHT-200198
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Glaucoma, Open-Angle
Keywords: open angle glaucoma; timolol; dorzolamide
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients with open angle glaucoma
  Interventions: Drug: Dorzolamide 2%
- 2 (Active Comparator): Patients with open angle glaucoma
  Interventions: Drug: Timolol 0.5%

INTERVENTIONS:
Drug: Dorzolamide 2%
  Arms: 1
Drug: Timolol 0.5%
  Arms: 2

SUMMARY:
Glaucoma is one of the most common causes of blindness in the industrialized nations. For a long time glaucoma has been defined as a disease in which high intraocular pressure (IOP) leads to irreversible optic disk damage and concommitant visual field loss. However, recent investigations show that IOP is not necessarily an adequate measure of clinical severity or a predictor of clinical progression: about 20% of all eyes with high IOP do not develop visual field loss and some patients suffering from visual field loss due to optic disk damage have normal IOP. Hence, factors other than IOP are likely involved in the pathogenesis of glaucoma. The role of vascular factors in the pathogenesis of glaucoma has recently received much attention and optic nerve head hypoperfusion may play a critical role in the development of glaucoma. It may therefore be important for an optimal prevention of visual field defects in glaucoma that the topical antiglaucoma drugs used do not only reduce IOP but also stabilize or enhance the perfusion of the optic nerve head.

Therefore, the aim of the present study is to compare the effect of a 3 months treatment with timolol or dorzolamide in patients with open angle glaucoma on optic disk blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 19 years
* Primary open angle glaucoma or ocular hypertension with IOP higher than 22 mmHg in at least one eye
* Washout period for previous antiglaucoma treatment: two weeks for adrenergic agonists, one week for parasympathomimetic agents

Exclusion Criteria:

* Exfoliation glaucoma, pigmentary glaucoma
* History of acute angle closure
* Intraocular surgery or argon laser trabeculoplasty within the last 6 months
* Ocular inflammation or infection within the last 3 months
* Contact lenses
* Patients with bradycardia (heart rate less than 50 beats/min)
* Second or third degree heart block
* Asthma
* COPD
* Congestive Heart Failure
* Severe renal impairment (Creatinine clearance less than 1.8 l/h
* History or hypersensitivity to one of the study drugs or drugs with similar chemical structure
* History of non-IOP responder to beta-blockers or carbonic anhydrase inhibitors
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 1999-05; Primary Completion 2001-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Percent change over baseline after 3 months of treatment of optic disk blood flow measured with the Heidelberg Retina Flowmeter | 5 minutes measurement of optic disk blood flow on 3 study days
Percent change over baseline after 3 months of treatment of fundus pulsation amplitude (FPA) in the optic disk as assessed with laser interferometry | 5 minutes measurement of FPA on 3 study days

CONTACTS AND LOCATIONS:
Overall Officials: Hans G Eichler, MD, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Fuchsjager-Mayrl G, Georgopoulos M, Hommer A, Weigert G, Pemp B, Vass C, Garhofer G, Schmetterer L. Effect of dorzolamide and timolol on ocular pressure: blood flow relationship in patients with primary open-angle glaucoma and ocular hypertension. Invest Ophthalmol Vis Sci. 2010 Mar;51(3):1289-96. doi: 10.1167/iovs.09-3827. Epub 2009 Oct 22. PMID 19850848